CLINICAL TRIAL: NCT04643626
Title: The Impact of Artificial Intelligence Dietary Smartphone Application on Nutritional Status Among Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: National Cancer Institute, Malaysia (Other Government)
Responsible Party: Principal Investigator, HO CHIOU YI, Principal Investigator, National Cancer Institute (NCI)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NMRR-19-2948-51031
Record Dates: First submitted 2020-11-03; First posted 2020-11-25 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Malnutrition, Calorie; Malnutrition; Protein; Weight Change, Body
Keywords: artificial intelligence dietary application; weight; oral intake
MeSH Terms: conditions — Malnutrition; Kwashiorkor; Body Weight Changes; Body Weight

STUDY DESIGN:
Intervention Model Description: Multi-center prospective pilot trial study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IG (Experimental): artificial intelligence dietary application, iDSA, will be introduced and installed. Explanation on the function and application of iDSA will be given. Daily energy and macro-nutrients requirement target will bed set. The daily energy and macronutrients requirement target is secured by password. Subjects will record their daily dietary intake (food with cooking method and portion size) and nutrition impact symptoms via smartphone application at least 3 times a week. Subjects able to keep track their intake at home. During follow up session, subjects show the iDSA diet intake summary records to Researcher for further assessment.
  Interventions: Device: artificial intelligence dietary android mobile application
- CG (No Intervention): CG will receive conventional dietitian care includes nutrition care process using conventional 24 hours diet recall method for dietary assessment

INTERVENTIONS:
Device: artificial intelligence dietary android mobile application — subjects use artificial intelligence dietary mobile application to monitor dietary intake
  Other Names: iDSA
  Arms: IG

SUMMARY:
Multi-center prospective pilot trial study

DETAILED DESCRIPTION:
This is a clinical study to evaluate impact of dietary smartphone application on nutritional status among cancer patients. the study hypotheses there is improvement in nutritional outcome in intervention group if compare with control group. the eligible subjects will be screened according to inclusion criteria and approached individually to participate in this study. The consented subjects will be divided randomly into two groups, intervention and conventional groups. Conventional dietitian care will be given to conventional group (CG) while intervention group (IG) will received innovated dietitian care where they will be introduced with iDSA apps and installed in consented subjects' smartphone. All subjects will be reviewed again by dietitian in 1-month time to assess nutritional status (weight and energy protein intake) as well as nutrition impact symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Possessing smartphone and is willing to use smartphone application
* Been referred to dietitian in outpatient clinic
* At least 18 years of age
* Malaysian

Exclusion Criteria:

* Inability to use the smartphone application (eg. due to vision problems)
* Not been referred to dietitian in outpatient clinic
* Patients who participate in other study at the same time
* On nutrition support (enteral / intra-venous)
* Vulnerable subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
weight changes | one month
  compare weight before intervention and after intervention
daily energy intake | one month
  compare daily energy intake before intervention and after intervention
daily protein intake | one month
  compare daily protein intake before intervention and after intervention

SECONDARY OUTCOMES:
PG-SGA score | one month
  compare PG-SGA score (numerical data) before intervention and after intervention
Nutrition Impact Symptoms (NIS) | one month
  compare NIS score (scale data) before intervention and after intervention. The score range from 1 to 5 where score 1 is better while score 5 is worst

CONTACTS AND LOCATIONS:
Overall Officials: Chiou Yi Ho, Principal Investigator — National Cancer Insitute, Malaysia
Locations (1):
- National Cancer Institute, Putrajaya, Putrajaya, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided